CLINICAL TRIAL: NCT06587672
Title: Factors Affecting Selection of Leadless Pacemaker in Patients with Atrioventricular Block and Atrioventricular Synchronous Pacing Status with a Micra AV: a Multicenter, Prospective, Observational Study
Brief Title: Factors Affecting Selection of Leadless Pacemaker and Atrioventricular Synchronous Pacing Status
Status: Not yet recruiting | Type: Observational
Sponsor: Xiaohan Fan (Other)
Collaborators: Tianjin Chest Hospital (Other); Beijing Friendship Hospital (Other); Beijing Hospital (Other Government); Peking University First Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaohan Fan, Professor, Fu Wai Hospital, Beijing, China
Organization: Fu Wai Hospital, Beijing, China (Other)
Other Study IDs: 2024-ZX028
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pacemaker; Atrioventricular Block; Clinical Trials; Pacing
Keywords: Leadless pacing; Atrioventricular synchrony; Atrioventricular block; Atrial contraction
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients received Micra AV implantation: Patients received Micra AV implantation
  Interventions: Device: Micra AV implantation

INTERVENTIONS:
Device: Micra AV implantation — Patients received Micra AV implantation

SUMMARY:
This is a multicenter, prospective, observational study ,the aim of this study is to find factors affecting selection of double-chamber leadless pacemaker in patients with atrioventricular block and ambulatory atrioventricular synchronous pacing status over time using a leadless ventricular pacemaker.

DETAILED DESCRIPTION:
Traditional pacemakers consist of a pulse generator and leads. Infections of the pulse generator pocket and lead-related complications are unavoidable issues in the application oftraditional pacemakers.Leadless pacemakers have emerged to address complications associated with the pacemaker pocket and leads in specific patients.The initial design of leadless pacemakers focused on single-chamber (right ventricular)sensing and pacing,However, patients with sinus rhythm may experience pacemakersyndrome symptoms due to atrioventricular desynchrony. Furthermore, a high proportion of atrioventricular dyssynchronous ventricular pacing might increase hospitalization rates for atrial fibrillation and heart failure.Recent developments in leadless dual-chamber pacemakersutilize a built-in triaxial accelerometer.This study aims to investigate factors considered by patients with atrioventricular block and clinical pacemaker implanting physicians when make sure the use of Micra AV. 2). It also seeks to evaluate the atrioventricular synchrony of Micra AV pacing in patients during both exercise and rest, while analyzing factors that influence the AV synchrony.For all screened patients, a questionnaire is required to be finished with data including age, gender, occupation, educational level, clinical history, comorbidities, previous infections, history of implanted electronic devices, economic status, and medical insurance conditions. At same time, all physicians are asked to complete a questionnaire for analyzing the factors influencing the decision of device option.An ambulatory electrocardiogram will be performed at 3 months, 6 months, and 1 year follow-up after device implantation. Data regarding the proportion of atrioventricular Research Protocol Template (Observational Study)_V1.0_2023.10.04 7/10 synchrony, atrial sensing atrial contraction mechanical wave (A4) threshold, ventricular pacing threshold, sensing, and impedance will be tested and collected. Postoperative exercise related symptoms and adverse events will be routinely tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with atrioventricular conduction block, meeting the indications for dual-chamber leadless pacemakers as per the "Chinese Expert Consensus on Clinical Application of Leadless Pacemakers (2022)".
2. Age ≥18 years.
3. Expected lifespan ≥1 year.
4. Consent to sign an informed consent form and cooperate in the collection of baseline data and subsequent follow-ups

Exclusion Criteria:

1. Patients anticipated to have a high ventricular pacing proportion (>40%) and with left ventricular ejection fraction less than 50%.
2. Patients with persistent atrial fibrillation and a high expected ventricular pacing proportion.
3. Post-tricuspid valve mechanical valve replacement surgery.
4. Patients with inferior vena cava pathway anomalies, precluding passage of the leadless pacemaker's delivery sheath.
5. Patients with an expected lifespan of less than 1 year. 6 Patients who are pregnant, planning pregnancy, or undergoing cardiac transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with atrioventricular conduction block, meeting the indications for dual-chamber leadless pacemakers as per the "Chinese Expert Consensus on Clinical Application of Leadless Pacemakers (2022)".All patients should sign written informed consent for agreement of the implantation procedure.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete the survey questionnair before implanting a pacemaker | 1 day before implanting a pacemaker
  Complete the survey questionnair
The percentage of atrioventricular synchrony at 3 months after Micra AV implantation. | 3 months post-implant
  The percentage of atrioventricular synchrony will be calculated based on the recording of a 20-minute resting period in the outpatient consulting room, via dividing the total number of AV synchronous cycles by the total number of cardiac cycles recoded by a Holter. An AV synchronous cycle will be defined as a paced or sensed ventricular beat within 300 ms following a surface ECG confirmed P-wave.

SECONDARY OUTCOMES:
Immediate success rate of Micra AV implantation. | During implantation on day 0
  Successfully implant a Micra AV during procedure.
The percentage of atrioventricular synchrony at 6, 12 months after Micra AV implantation. | 6, 12 months post-implant
  The percentage of atrioventricular synchrony will be calculated based on the recording of a 20-minute resting period in the outpatient consulting room, via dividing the total number of AV synchronous cycles by the total number of cardiac cycles recoded by a Holter. An AV synchronous cycle will be defined as a paced or sensed ventricular beat within 300 ms following a surface ECG confirmed P-wave.
Ventricular pacing threshold, at 3 months, 6 months, and 1 year after Micra AV implantation. | 3, 6, 12months post-implant
  Measuring the ventricular pacing threshold by a programmer at the outpatient clinic at 3,6 and 12 month.
Ventricular sensing at 3 months, 6 months, and 1 year after Micra AV implantation. | 3, 6, 12 months post-implant
  Measuring ventricular sensing by a programmer at the outpatient clinic at 3,6 and 12 month.
Impedance at 3 months, 6months, and 1 year after Micra AV implantation. | 3, 6, 12 months post-implant
  Measuring Impedance by a programmer at the outpatient clinic at 3,6 and 12 month.
Major complications related to the device implantation at perioperative period, and 3, 6, 9, 12 months after Micra AV implantation | Days 0,1 and 3, 6, 9, 12 months post- implant
  Major complations related to the device implantation include, pericardial effusion, dislodgement, threshold elevation or loss of capture, infection, etc.
All-cause mortality rates at 3 months, 6 months, and 1 year after Micra AV implantation. | 3, 6, 9, 12 months post-implant
  These data will be collected at the outpatient clinic at 3,6 and 12 month, 9-month follow-up will be conducted via telephone.
Rehospitalization events related to heart failure at 3 months, 6 months, and 1year after Micra AV implantation. | 3, 6, 12 months post-implant
  Rehospitalization events due to heart failure at 3 months, 6 months, and 1year after Micra AV implantation.
Tachycardia related to the pacemaker, or adverse events related to the device or algorithm at 3, 6, 12 months after Micra AV implantation. | 3,6,12 months post-implant
  Tachycardia or or adverse events related to the device or algorithm during the follow-up
Left venriculat ejection fraction measured by echocardiography at 6, 12 months after Micra AV implanted | 6, 12 months post-implant
  Left venriculat ejection fraction measured by echocardiography.
Left ventricular end-diastolic diameter measured by echocardiography at 6, 12 months after Micra AV implantation. | 6, 12 months post-implant
  Left ventricular end-diastolic diameter measured by echocardiography
Parameter adjustment events related to the synchrony less than 70% at 3, 6, 12 months after Micra AV implantation.. | 3, 6, 12months post-implant
  Parameter adjustment event will be defined as optimamizing the pacemaker parameters due to synchrony less than 70%.
Arrhythmias events at 3, 6, 12 months after Micra AV implantion | 3, 6, 12months post-implant
  All kinds of arrhythmias events recorded via electrocardiogram or device during the follow up
Syncope events at 3, 6, 12 months after Micra AV implantion | 3, 6, 12months post-implant
  Syncope events during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan Fan, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - Fu Wai Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ann HW, Ahn JY, Jeon YD, Jung IY, Jeong SJ, Joung B, Lee M, Ku NS, Han SH, Kim JM, Choi JY. Incidence of and risk factors for infectious complications in patients with cardiac device implantation. Int J Infect Dis. 2015 Jul;36:9-14. doi: 10.1016/j.ijid.2015.05.011. Epub 2015 May 14. PMID 25980618
- [Background] Wilkoff BL. How to treat and identify device infections. Heart Rhythm. 2007 Nov;4(11):1467-70. doi: 10.1016/j.hrthm.2007.08.007. Epub 2007 Aug 11. No abstract available. PMID 17954409
- [Background] Johansen JB, Jorgensen OD, Moller M, Arnsbo P, Mortensen PT, Nielsen JC. Infection after pacemaker implantation: infection rates and risk factors associated with infection in a population-based cohort study of 46299 consecutive patients. Eur Heart J. 2011 Apr;32(8):991-8. doi: 10.1093/eurheartj/ehq497. Epub 2011 Jan 20. PMID 21252172
- [Background] Knops RE, Tjong FV, Neuzil P, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Reddy VY. Chronic performance of a leadless cardiac pacemaker: 1-year follow-up of the LEADLESS trial. J Am Coll Cardiol. 2015 Apr 21;65(15):1497-504. doi: 10.1016/j.jacc.2015.02.022. PMID 25881930
- [Background] Reddy VY, Knops RE, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Tjong FV, Jacobson P, Ostrosff A, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Neuzil P. Permanent leadless cardiac pacing: results of the LEADLESS trial. Circulation. 2014 Apr 8;129(14):1466-71. doi: 10.1161/CIRCULATIONAHA.113.006987. Epub 2014 Mar 24. PMID 24664277
- [Background] Reynolds DW, Ritter P. A Leadless Intracardiac Transcatheter Pacing System. N Engl J Med. 2016 Jun 30;374(26):2604-5. doi: 10.1056/NEJMc1604852. No abstract available. PMID 27355552